CLINICAL TRIAL: NCT04696367
Title: Impact of Nutritional Deficit in Emergency Surgery: A Pilot Study
Brief Title: Impact of Nutritional Deficit in Emergency Surgery
Acronym: INDIcatES
Status: Completed | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: STH20936
Record Dates: First submitted 2019-12-10; First posted 2021-01-06 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Emergencies; Surgery; Malnutrition
Keywords: emergency surgery; malnutrition; pilot study
MeSH Terms: conditions — Emergencies; Malnutrition | interventions — Laparotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with acute intra-abdominal pathology: Patients admitted to hospital with acute intra-abdominal pathology
  Interventions: Procedure: Emergency laparotomy

INTERVENTIONS:
Procedure: Emergency laparotomy — Midline laparotomy for acute intra-abdominal pathology
  Other Names: Celiotomy

SUMMARY:
Patients in emergency settings might become malnourished. There are different ways to identify the group as 'at risk' of malnutrition. There are also several different ways to measure outcomes. This pilot study will look at patients undergoing emergency laparotomy, investigate relationships between different selection criteria and outcome measures, and test feasibility of outcome measure collection.

DETAILED DESCRIPTION:
Patients in emergency settings might become malnourished. There are different ways to identify the group as 'at risk' of malnutrition. There are also several different ways to measure outcomes. This pilot study will look at patients undergoing emergency laparotomy, investigate relationships between different selection criteria and outcome measures, and test feasibility of outcome measure collection.

ELIGIBILITY:
Inclusion Criteria:

* Willing to consent,

  -≥ 18 years old
* eligible for inclusion in National Emergency Laparotomy Audit
* first procedure during admission (<7 days from admission).

Exclusion Criteria:

* Recent discharge from hospital (within 60 days),
* unable to provide informed consent
* life expectancy <12 months
* prisoners
* lack mental capacity
* language barrier affecting ability to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending two UK hospitals which provide emergency surgery services who require an emergency laparotomy
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Time without nutrition (measured in days) | within 90 days of admission to hospital
  This is defined as the time elapsed between last normal enteral intake, and resumption of enteral intake, or naso-enteric feeding, or parenteral nutrition.

SECONDARY OUTCOMES:
In hospital complications | within 90 days of admission to hospital
  Complications related to surgery measured using the comprehensive complication index
Feasibility of completion of complications at day of discharge | within 90 days of admission to hospital
  Proportion of patients with a completed comprehensive complication index
Change in health utility | Measurements take at baseline, 5 days post-operatively and 90 days post-operatively
  Measured using EQ-5D-5L (EuroQol- five dimension - five level)
Feasibility of completion of EQ-5D-5L (EuroQol- five dimension - five level) at 90 days | 90 days post operatively
  Reported as proportion of respondents replying

CONTACTS AND LOCATIONS:
Overall Officials: Timothy O'Connor, MBChB, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Doncaster Royal Infirmary, Doncaster, South Yorkshire
  - Sheffield Teaching Hospitals, Sheffield, South Yorkshire

IPD SHARING:
Plan to Share IPD: No